CLINICAL TRIAL: NCT00360529
Title: A Twenty Four Week, Randomized, Double-Blind, Placebo-Controlled, Safety and Efficacy Trial of Flibanserin 50mg Every Evening and Flibanserin 100mg Every Evening in Women With Hypoactive Sexual Desire Disorder in North America
Brief Title: 24-week Placebo-controlled Trial of Flibanserin Once Daily in Premenopausal Women With Hypoactive Sexual Desire Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sprout Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 511.71; VIOLET (Other Grant/Funding Number: Boehringer Ingelheim)
Record Dates: First submitted 2006-08-03; First posted 2006-08-04 (Estimated); Results first posted 2016-06-27 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-06

CONDITIONS: Sexual Dysfunctions, Psychological
MeSH Terms: conditions — Sexual Dysfunctions, Psychological | interventions — flibanserin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- fibanserin (Experimental): flibanserin 50 mg q.h.s.
  Interventions: Drug: flibanserin
- flibanserin (Experimental): flibanserin 100 mg q.h.s.
  Interventions: Drug: flibanserin
- placebo (Placebo Comparator): placebo q.h.s.
  Interventions: Drug: flibanserin

INTERVENTIONS:
Drug: flibanserin — flibanserin placebo versus 50 mg qhs versus 100 mg qhs
  Other Names: flibanserin 50 mg; flibanserin 100mg; placebo

SUMMARY:
This trial is designed to assess the safety and efficacy of flibanserin in the treatment of premenopausal women with Hypoactive Sexual Desire Disorder (HSDD) that meets standard diagnostic criteria. Efficacy for flibanserin will be assessed vs. a parallel placebo group.

DETAILED DESCRIPTION:
This trial was designed as a prospective, multicenter trial containing a 24-week, randomized, double blind, placebo controlled, parallel-group period that assessed the effects of flibanserin (maximum total daily dose: 100 mg q.d.) compared with placebo in premenopausal women with HSDD, determined by Diagnostic and Statistical Manual IV- Text Revision (DSM IV-TR®) criteria. Three hundred patients were to be randomized to each treatment group. This trial examined the safety and efficacy of flibanserin compared to placebo for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Women who are 18 years of age and older.
2. Premenopausal women having regular menstrual periods who have HSDD (decreased sexual desire), generalized acquired type, according to DSM IV-TR criteria.
3. Patient must meet minimum cut-off scores on questionnaires relating to sexual functioning and sexual distress.
4. Patients must be willing to try to have sexual activity (e.g., any act involving direct genital stimulation) at least once monthly.
5. Patients must be willing and able to use an electronic diary (eDiary) on a daily basis (e.g., have access to a working land line telephone for daily data transmissions).
6. At the Baseline Visit, patients must have complied with eDiary use adequately.
7. Patients must be in a stable, monogamous, heterosexual relationship that is secure and communicative, for at least 1 year prior to the Screen Visit. The partner is expected to be physically present at least 50% of each month.
8. Patients must have used a medically acceptable method of contraception for at least 3 months before the Baseline Visit (Visit 2) and continue to use that medically acceptable method of contraception during the trial.
9. In the investigators opinion, patients must be reliable, honest, compliant, and agree to co-operate with all trial evaluations as well as to be able to perform them.
10. Patients must be able and willing to give meaningful, written informed consent prior to participation in the trial, in accordance with regulatory requirements. Patients must have sufficient understanding to communicate effectively with the investigator, and be willing to discuss their sexual functioning with the investigative staff.
11. Patients must have a clinically acceptable Pap smear as read by a cytology facility (no evidence of malignancy or squamous intraepithelial lesions) within 6 months before the Screen Visit.

Exclusion Criteria:

1. Patients who have taken any medication noted in the protocols List of Prohibited Medications within 30 days before screening.
2. Patients whose sexual function was affected (enhanced or worsened) in the investigators opinion by any medication within 30 days before the Screen Visit and anytime prior to the Baseline Visit.
3. Patients with a history of drug dependence or abuse within the past one year.
4. Patients with a history of multiple severe reactions (i.e., allergic or oversensitivity to usual doses) to drugs that affect the brain.
5. Patients with a history of participation in a trial of another investigational medication within one month prior to the Screen Visit, or participation in any previous clinical trial of flibanserin.
6. Patients who meet accepted diagnostic criteria for sexual disorders that would interfere with improvement in HSDD (sexual aversion, substance-induced sexual problems, urge to live as a man, etc.
7. Patients who indicate that their sexual partner has inadequately treated sexual problems that could interfere with the patients response to treatment.
8. Patients who have entered the menopausal transition or menopause or have had a hysterectomy.
9. Patients with findings at the Screen Visit of infection, inflammation, undue tenderness, or shrinkage (atrophy) of the female organs.
10. Patients who are breast feeding or have breastfed within the last 6 months prior to the Baseline Visit.
11. Patients who are pregnant or have been pregnant within the last 6 months prior to the Baseline Visit.
12. Patients with a history of Major Depressive Disorder within 6 months prior the Screen Visit, a score indicating depression on a depression scale, a history of suicide attempt, or current suicidal ideation evident at the Screen or Baseline Visit.
13. Patients with a history of any other psychiatric disorders that could impact sexual function, risks patients safety, or may impact compliance.

<truncated>

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 880 (Actual)
Dates: Start 2006-07; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sprout Pharmaceuticals, Study Chair — Sprout Pharmaceuticals
Locations (54):
- United States (40):
  - 511.71.01034 Boehringer Ingelheim Investigational Site, Mobile, Alabama
  - 511.71.01042 Boehringer Ingelheim Investigational Site, South Birmingham, Alabama
  - 511.71.01016 Boehringer Ingelheim Investigational Site, Phoenix, Arizona
  - 511.71.01041 Boehringer Ingelheim Investigational Site, La Mesa, California
  - 511.71.01011 Boehringer Ingelheim Investigational Site, San Diego, California
  - 511.71.01027 Boehringer Ingelheim Investigational Site, Westlake Village, California
  - 511.71.01035 Boehringer Ingelheim Investigational Site, Denver, Colorado
  - 511.71.01010 Boehringer Ingelheim Investigational Site, Groton, Connecticut
  - 511.71.01021 Boehringer Ingelheim Investigational Site, New Britain, Connecticut
  - 511.71.01037 Boehringer Ingelheim Investigational Site, Newark, Delaware
  - 511.71.01001 Boehringer Ingelheim Investigational Site, Boynton Beach, Florida
  - 511.71.01032 Boehringer Ingelheim Investigational Site, Clearwater, Florida
  - 511.71.01014 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 511.71.01025 Boehringer Ingelheim Investigational Site, Pembroke Pines, Florida
  - 511.71.01006 Boehringer Ingelheim Investigational Site, Plantation, Florida
  - 511.71.01015 Boehringer Ingelheim Investigational Site, Atlanta, Georgia
  - 511.71.01038 Boehringer Ingelheim Investigational Site, Marietta, Georgia
  - 511.71.01036 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 511.71.01029 Boehringer Ingelheim Investigational Site, Evansville, Indiana
  - 511.71.01028 Boehringer Ingelheim Investigational Site, Renton, Indiana
  - 511.71.01024 Boehringer Ingelheim Investigational Site, New Orlean, Louisiana
  - 511.71.01040 Boehringer Ingelheim Investigational Site, Towson, Maryland
  - 511.71.01045 Boehringer Ingelheim Investigational Site, Brighton, Massachusetts
  - 511.71.01005 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 511.71.01030 Boehringer Ingelheim Investigational Site, Albuquerque, New Mexico
  - 511.71.01007 Boehringer Ingelheim Investigational Site, Rochester, New York
  - 511.71.01012 Boehringer Ingelheim Investigational Site, The Bronx, New York
  - 511.71.01023 Boehringer Ingelheim Investigational Site, New Bern, North Carolina
  - 511.71.01002 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 511.71.01044 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 511.71.01026 Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - 511.71.01039 Boehringer Ingelheim Investigational Site, Edmond, Oklahoma
  - 511.71.01003 Boehringer Ingelheim Investigational Site, Danville, Pennsylvania
  - 511.71.01033 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 511.71.01031 Boehringer Ingelheim Investigational Site, Pittsburgh, Pennsylvania
  - 511.71.01022 Boehringer Ingelheim Investigational Site, Mt. Pleasant, South Carolina
  - 511.71.01020 Boehringer Ingelheim Investigational Site, Germantown, Tennessee
  - 511.71.01017 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 511.71.01018 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 511.71.01008 Boehringer Ingelheim Investigational Site, Huntington, West Virginia
- Canada (14):
  - 511.71.02002 Boehringer Ingelheim Investigational Site, Calgary, Alberta
  - 511.71.02006 Boehringer Ingelheim Investigational Site, Kelowna, British Columbia
  - 511.71.02011 Boehringer Ingelheim Investigational Site, Surrey, British Columbia
  - 511.71.02007 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 511.71.02008 Boehringer Ingelheim Investigational Site, Victoria, British Columbia
  - 511.71.02012 Boehringer Ingelheim Investigational Site, Victoria, British Columbia
  - 511.71.02010 Boehringer Ingelheim Investigational Site, Winnipeg, Manitoba
  - 511.71.02001 Boehringer Ingelheim Investigational Site, Halifax, Nova Scotia
  - 511.71.02004 Boehringer Ingelheim Investigational Site, Burlington, Ontario
  - 511.71.02013 Boehringer Ingelheim Investigational Site, London, Ontario
  - 511.71.02009 Boehringer Ingelheim Investigational Site, Oshawa, Ontario
  - 511.71.02003 Boehringer Ingelheim Investigational Site, Ottawa, Ontario
  - 511.71.02005 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 511.71.02014 Boehringer Ingelheim Investigational Site, Québec, Quebec

REFERENCES:
- [Derived] Derogatis LR, Komer L, Katz M, Moreau M, Kimura T, Garcia M Jr, Wunderlich G, Pyke R; VIOLET Trial Investigators. Treatment of hypoactive sexual desire disorder in premenopausal women: efficacy of flibanserin in the VIOLET Study. J Sex Med. 2012 Apr;9(4):1074-85. doi: 10.1111/j.1743-6109.2011.02626.x. Epub 2012 Jan 16. PMID 22248038

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: placebo at bedtime
- Flibanserin 50 mg q.h.s.: Flibanserin 50 mg at bedtime
- Flibanserin 100 mg q.h.s: Flibanserin 100 mg at bedtime
Period: Overall Study
Arm/Group | Placebo | Flibanserin 50 mg q.h.s. | Flibanserin 100 mg q.h.s
Started | 295 | 295 | 290
Completed | 234 | 230 | 199
Not Completed | 61 | 65 | 91
Not completed — Adverse Event | 10 | 23 | 33
Not completed — Protocol Violation | 3 | 3 | 11
Not completed — Lost to Follow-up | 14 | 10 | 13
Not completed — Withdrawal by Subject | 22 | 14 | 18
Not completed — Lack of Efficacy | 8 | 6 | 5
Not completed — Reason discontinued not explained above | 4 | 9 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Flibanserin 50 mg q.h.s. | Flibanserin 100 mg q.h.s | Total
Number analyzed (Participants) | 295 | 295 | 290 | 880
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.5 (7.0) | 36.3 (7.5) | 35.6 (7.2) | 35.8 (7.2)
Age, Customized [Number; unit: participants]
  18 - 34 years | 126 | 127 | 134 | 387
  35 - 44 years | 136 | 125 | 118 | 379
  >= 45 years | 33 | 43 | 38 | 114
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 295 | 295 | 290 | 880
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 235 | 237 | 229 | 701
  White Hispanic | 21 | 26 | 19 | 66
  Black Hispanic | 2 | 1 | 1 | 4
  Black | 31 | 29 | 35 | 95
  Asian | 6 | 2 | 4 | 12
  Asian Hispanic | 0 | 0 | 1 | 1
  Missing | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 66 | 69 | 66 | 201
  United States | 229 | 226 | 224 | 679
Marital Status [Number; unit: participants]
  Unmarried | 58 | 81 | 61 | 200
  Married | 237 | 214 | 229 | 680
Education level [Number; unit: participants]
  Partial high school | 1 | 6 | 3 | 10
  High school graduate or equivalent | 35 | 33 | 26 | 94
  Partial college/university | 78 | 80 | 85 | 243
  College/university graduate | 139 | 131 | 130 | 400
  Post-graduate/professional degree | 42 | 45 | 46 | 133
  Missing | 0 | 0 | 0 | 0
Employment status [Number; unit: participants]
  Full time (>= 40 hours/week) | 195 | 194 | 180 | 569
  Part time (17-39 hours/week) | 54 | 58 | 48 | 160
  Occassional (1-16 hours/week) | 5 | 8 | 15 | 28
  Full time homemaker | 33 | 28 | 31 | 92
  Unemployed | 8 | 7 | 16 | 31
  Missing | 0 | 0 | 0 | 0
How long in present relationship [Mean (Standard Deviation); unit: years] | 10.39 (6.50) | 11.05 (6.94) | 10.48 (6.38) | 10.64 (6.61)
Alcohol status [Number; unit: participants]
  Non drinker | 68 | 83 | 78 | 229
  Drinks - no interference | 227 | 212 | 212 | 651
  Drinks - possible interference | 0 | 0 | 0 | 0
Smoking history [Number; unit: participants]
  Never smoked | 200 | 202 | 206 | 608
  Ex-smoker | 60 | 56 | 55 | 171
  Currently smokes | 35 | 37 | 29 | 101
Smoking history - pack years [Mean (Standard Deviation); unit: pack years] | 6.72 (7.27) | 6.46 (6.09) | 6.07 (8.26) | 6.43 (7.20)
Weight [Mean (Standard Deviation); unit: kilograms] | 71.09 (15.31) | 72.78 (17.05) | 74.19 (17.53) | 72.68 (16.68)
Body mass index [Mean (Standard Deviation); unit: kilogram/square meter] | 26.35 (6.07) | 26.90 (6.13) | 27.04 (5.85) | 26.76 (6.02)

OUTCOME MEASURES:

1. Primary Outcome: Satisfying Sexual Event Monthly Change From Baseline at Final Visit
Description: Change from baseline in the frequency of sexual satisfying events, as measured via e-Diary, standardized to a 28-day period. Change from baseline is calculated as the difference between the four week baseline period and Week 21 to Week 24.
Time Frame: Baseline, Week 24
Population: The Full Analysis Set (FAS) consisted of those patients who were randomized to a treatment group, received at least one dose of study medication, and had at least one on-treatment efficacy assessment. The FAS was analyzed for efficacy.
Measure: Mean (Standard Deviation); unit: number of events
Arm/Group | Placebo | Flibanserin 50 mg q.h.s. | Flibanserin 100 mg q.h.s
Number analyzed (Participants) | 285 | 291 | 275
number of events | 0.8 (3.4) | 1.4 (3.6) | 1.6 (3.8)
Statistical Analysis 1: Comparison: Placebo vs Flibanserin 50 mg q.h.s; Flibanserin 50 mg qhs versus placebo; Test type: Superiority or Other; p = 0.0454, Wilcoxon (Mann-Whitney) — Hierarchical ordering used for multiple endpoints, and Hochberg used for multiple dose comparisons. P-values ordered (p1≤p2). If p2≤0.05 then all doses significant. If p1≤0.025 then reject null for p1
Statistical Analysis 2: Comparison: Placebo vs Flibanserin 100 mg q.h.s; Flibanserin 100 mg qhs versus placebo; Test type: Superiority or Other; p = 0.0024, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

2. Primary Outcome: Sexual Desire Monthly Change on Electronic Diary From Baseline at Final Visit
Description: Change from baseline in eDiary Sexual Desire Monthly Total Score standardized to a 28-day period. Change from baseline calculated as the difference between the 4 week baseline period and Week 21 to Week 24. Patients recorded information daily throughout trial. Every time the eDiary was completed, a desire question was asked. If a patient did not complete the diary on a given day, the patient was not asked to enter desire information for more than a 24-hour retrospective period. The desire item read "Indicate your most intense level of sexual desire in the last 24 hours/since your last visit." Potential responses included "no," "low," "moderate," or "strong", scored 0-3 (0 indicating no desire and 3 indicating the highest level of desire):
  0 = No desire
  1. = Low desire
  2. = Moderate desire
  3. = Strong desire
  Total score ranged from 0-84, with higher scores reflecting stronger desire). Monthly desire score was calculated as 28 x (sum of daily desire scores/number of responses).
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Flibanserin 50 mg q.h.s. | Flibanserin 100 mg q.h.s
Number analyzed (Participants) | 285 | 291 | 275
units on a scale | 6.9 (0.9) | 8.2 (0.9) | 9.1 (1.0)
Statistical Analysis 1: Comparison: Placebo vs Flibanserin 50 mg q.h.s; Flibanserin 50 mg qhs versus placebo; Test type: Superiority or Other; p = 0.2606, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Model includes treatment, centre and baseline as a covariate; Mean Difference (Final Values) = 1.3, 95% CI [-1.0 to 3.7]
Statistical Analysis 2: Comparison: Placebo vs Flibanserin 100 mg q.h.s; Flibanserin 100 mg qhs versus placebo; Test type: Superiority or Other; p = 0.066, ANCOVA; Model includes treatment, centre and baseline as a covariate; Mean Difference (Final Values) = 2.2, 95% CI [-0.1 to 4.6]

3. Secondary Outcome: Female Sexual Distress Scale - Revised (FSDS-R) Total Score Change From Baseline at Final Visit
Description: Change from baseline in the Female Sexual Distress Scale - revised (FSDS-R) Total Score with a seven day recall period.
  The FSDS is a measure of female personal distress associated with sexual dysfunction. Reliability and validity of the FSDS (12-item version) has been evaluated in different samples of sexually functional and dysfunctional women. An additional question (Question 13) was added to the validated FSDS© in order to capture distress related to specifically sexual desire so that this domain could be appropriately captured. FSDS plus Question 13 comprises FSDS-R, thus making the FSDS-R a self-administered 13 item questionnaire. The maximum total score of the FSDS-R is '52' (score of minimum of 0 and maximum of 4 for each item) and indicates the maximum level of sexual distress (the higher the score, the higher the level of reported sexual desire).
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Flibanserin 50 mg q.h.s. | Flibanserin 100 mg q.h.s
Number analyzed (Participants) | 289 | 293 | 280
score on a scale | -4.9 (0.7) | -6.1 (0.7) | -8.9 (0.7)
Statistical Analysis 1: Comparison: Placebo vs Flibanserin 50 mg q.h.s; Flibanserin 50 mg qhs versus placebo; Test type: Superiority or Other; p = 0.1601, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Model includes treatment, centre and baseline as a covariate; Mean Difference (Final Values) = -1.2, 95% CI [-2.9 to 0.5]
Statistical Analysis 2: Comparison: Placebo vs Flibanserin 100 mg q.h.s; Flibanserin 100 mg qhs versus placebo; Test type: Superiority or Other; p = 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Model includes treatment, centre and baseline as a covariate; Mean Difference (Final Values) = -3.9, 95% CI [-5.6 to -2.2]

4. Secondary Outcome: Female Sexual Distress Scale - Revised (FSDS-R) Question 13 Score Change From Baseline at Final Visit
Description: Change from baseline in the FSDS-R Question 13 (Bothered by low sexual desire). The FSDS is a measure of female personal distress associated with sexual dysfunction. Reliability and validity of the FSDS (12-item version) has been evaluated in different samples of sexually functional and dysfunctional women. An additional question (Question 13) was added to the validated FSDS© in order to capture distress related to specifically sexual desire so that this domain could be appropriately captured. FSDS plus Question 13 comprises FSDS-R, thus making the FSDS-R a self-administered 13 item questionnaire. The scoring for item 13 is from 0-4, with 4 indicating the highest level of sexual distress.
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Flibanserin 50 mg q.h.s. | Flibanserin 100 mg q.h.s
Number analyzed (Participants) | 289 | 293 | 280
score on a scale | -0.5 (0.1) | -0.6 (0.1) | -0.8 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Flibanserin 50 mg q.h.s; Flibanserin 50 mg qhs versus placebo; Test type: Superiority or Other; p = 0.1144, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Model includes treatment, centre and baseline as a covariate; Mean Difference (Final Values) = -0.1, 95% CI [-0.3 to 0.0]
Statistical Analysis 2: Comparison: Placebo vs Flibanserin 100 mg q.h.s; Flibanserin 100 mg qhs versus placebo; Test type: Superiority or Other; p = 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Model includes treatment, centre and baseline as a covariate; Mean Difference (Final Values) = -0.4, 95% CI [-0.5 to -0.2]

5. Secondary Outcome: Female Sexual Functioning Index (FSFI) Desire Domain Score Change From Baseline at Final Visit
Description: Female Sexual Function Inventory (FSFI) Desire Domain assesses sexual desire or interest with 2 questions ranging from 1 (very low) to 5 (very high). The domain total score is multiplied by 0.6 yielding scores ranging from 1.2 to 6 (higher scores = higher level of desire or interest).
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Flibanserin 50 mg q.h.s. | Flibanserin 100 mg q.h.s
Number analyzed (Participants) | 290 | 293 | 280
score on a scale | 0.5 (0.1) | 0.8 (0.1) | 0.9 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Flibanserin 50 mg q.h.s; Flibanserin 50 mg qhs versus placebo; Test type: Superiority or Other; p = 0.0173, ANCOVA; Model includes treatment, centre and baseline as a covariate; Mean Difference (Final Values) = 0.2, 95% CI [0.0 to 0.4]
Statistical Analysis 2: Comparison: Placebo vs Flibanserin 100 mg q.h.s; Flibanserin 100 mg qhs versus placebo; Test type: Superiority or Other; p = 0.0001, ANCOVA; Model includes treatment, centre and baseline as a covariate; Mean Difference (Final Values) = 0.4, 95% CI [0.2 to 0.5]

6. Secondary Outcome: Female Sexual Functioning Index (FSFI) Total Score Change From Baseline at Final Visit
Description: The FSFI© is a self-administered questionnaire to assess FSD, which consists of 19 questions that are scored from '0' to '5.' The scale contains six domains: desire, arousal, lubrication, orgasm, satisfaction, and pain. Higher scores indicate higher levels of the domain assessed. The total score is a weighted average of the six domains, each contributing a maximum of 6 points to the total, so the minimum score is 2, while the maximum score of FSFI© is 36.
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Flibanserin 50 mg q.h.s. | Flibanserin 100 mg q.h.s
Number analyzed (Participants) | 289 | 292 | 280
score on a scale | 2.4 (0.4) | 3.9 (0.4) | 5.0 (0.4)
Statistical Analysis 1: Comparison: Placebo vs Flibanserin 50 mg q.h.s; Flibanserin 50 mg qhs versus placebo; Test type: Superiority or Other; p = 0.0071, ANCOVA; Model includes treatment, centre and baseline as a covariate; Mean Difference (Final Values) = 1.5, 95% CI [0.4 to 2.6]
Statistical Analysis 2: Comparison: Placebo vs Flibanserin 100 mg q.h.s; Flibanserin 100 mg qhs versus placebo; Test type: Superiority or Other; p = 0.0001, ANCOVA; Model includes treatment, centre and baseline as a covariate; Mean Difference (Final Values) = 2.5, 95% CI [1.4 to 3.6]

7. Secondary Outcome: Patient Benefit Evaluation
Description: The Patient Benefit Evaluation is a single question asking the patient whether or not she experienced a meaningful benefit from the study medication during the trial. This question ("Overall, do you believe that you have experienced a meaningful benefit from the study medication?") was asked upon treatment discontinuation.
Time Frame: Week 24
Population: This question was asked at Week 24 only, so did not include participants who had discontinued the trial prior to that time (e.g., analysis population includes treatment completers only).
Measure: Number; unit: participants
Arm/Group | Placebo | Flibanserin 50 mg q.h.s. | Flibanserin 100 mg q.h.s
Number analyzed (Participants) | 266 | 271 | 254
participants
  Meaningful benefit from medication | 71 | 94 | 98
  No meaningful benefit from medication | 195 | 177 | 156
Statistical Analysis 1: Comparison: Placebo; Flibanserin 25 mg bid versus placebo; Test type: Superiority or Other; p = 0.0513, Cochran-Mantel-Haenszel; Model includes treatment and centre; Percentage responders = 34.7, 95% CI [29.0 to 40.4]
Statistical Analysis 2: Comparison: Placebo vs Flibanserin 50 mg q.h.s; Flibanserin 50 mg qhs versus placebo; Test type: Superiority or Other; p = 0.0059, Cochran-Mantel-Haenszel; Model includes treatment and centre; Percentage responders = 38.6, 95% CI [32.6 to 44.6]

ADVERSE EVENTS:
Arm/Group | Placebo | Flibanserin 50 mg q.h.s. | Flibanserin 100 mg q.h.s
Serious Adverse Events (participants affected / at risk) | 0/295 | 2/295 | 3/290
Other Adverse Events (participants affected / at risk) | 87/295 | 107/295 | 135/290
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=295) | Flibanserin 50 mg q.h.s. (N=295) | Flibanserin 100 mg q.h.s (N=290)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=295) | Flibanserin 50 mg q.h.s. (N=295) | Flibanserin 100 mg q.h.s (N=290)
Nausea (Gastrointestinal disorders) | 12 (12) | 23 (23) | 33 (33)
Fatigue (General disorders) | 8 (8) | 10 (10) | 18 (18)
Nasopharyngitis (Infections and infestations) | 24 (24) | 26 (26) | 18 (18)
Sinusitis (Infections and infestations) | 9 (9) | 7 (7) | 18 (18)
Upper respiratory tract infection (Infections and infestations) | 15 (15) | 22 (22) | 13 (13)
Dizziness (Nervous system disorders) | 5 (5) | 15 (15) | 26 (26)
Headache (Nervous system disorders) | 27 (27) | 22 (27) | 22 (22)
Somnolence (Nervous system disorders) | 9 (9) | 26 (26) | 32 (32)
Insomnia (Psychiatric disorders) | 16 (16) | 5 (5) | 21 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Sprout Pharmaceuticals publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract